CLINICAL TRIAL: NCT05197608
Title: At-risk and vulNerable Individuals To Infection With COVID-19 and ProActive inTervention With intEgrated Health and Social Care (ANTICIPATE): a Pragmatic Randomized Controlled Trial
Brief Title: At-risk and vulNerable Individuals To Infection With COVID-19 and ProActive inTervention With intEgrated Health and Social Care
Acronym: ANTICIPATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Ontario Medical Association (Other); Platinum Medical Clinic (Unknown); Markham Family Health Team (Unknown); Barrie and Community Family Health Team (Unknown); University of Toronto Practice Based Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SMH 20-140
Record Dates: First submitted 2021-09-27; First posted 2022-01-19 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Emotional Distress; Quality of Life; Mental Health
Keywords: Social Determinants of Health; COVID-19; primary health care; proactive care
MeSH Terms: conditions — Psychological Well-Being; COVID-19

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into "intervention" or "control" group.
  The intervention group will be connected to a system navigator who is a trained staff member embedded within the primary health clinic team with a focus to address participant's biological, psychological and social needs. Control group will be provided a tailored list of community resources.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - System Navigator (Experimental): The intervention group will be connected to a system navigator who is a trained staff member embedded within the primary health clinic team with a focus to address participant's biological, psychological and social needs.
  Working with the System Navigator will mean:
  * Discussing patients' current health status and concerns
  * Receiving support on management of chronic diseases and mental health including connection to local resources e.g. counseling, harm reduction, crisis support services
  * Receiving information about benefits that they may be entitled to and learning about free services
  * Receiving help from the System Navigator on forms or letters that are required to access resources
  Interventions: Other: System Navigator
- Tailored list of community resources (Active Comparator): Control group will be provided a tailored list of community resources.
  Interventions: Other: Tailored list of resources

INTERVENTIONS:
Other: System Navigator — Participants will be connected to a System Navigator, who is a trained staff embedded within their primary health clinic to support and help navigate biological, psychological and social needs in proactively identified vulnerable patients.
  Arms: Intervention - System Navigator
Other: Tailored list of resources — Control group will be provided a tailored list of resources
  Arms: Tailored list of community resources

SUMMARY:
This randomized control trial aims to explore a data-driven, proactive approach to identifying patients at greatest risk during the pandemic, and assess the impact of an embedded System Navigator in a primary health care setting. The System Navigator works one-on-one with patients to identify and provide support to their biological, psychological and social needs (e.g. income, housing, food security). Investigators are doing this study to find out whether proactive identification of vulnerable patients and linking to a System Navigator leads to reduction in emotional distress associated with managing complex health conditions and unmet social needs during COVID-19, compared to usual care.

Investigators will involve approximately 180 patients from primary care clinics that are a part of the University of Toronto Practice-Based Research Network (UTOPIAN). The information from this study will be used to help us understand how proactive engagement within a primary health setting can help to improve the health of patients during COVID-19, and beyond.

ELIGIBILITY:
Inclusion Criteria:

* At-risk and vulnerable patients of primary care organizations who are 60+ AND have one or more of:

  1. chronic condition (diabetes, CHF, CAD, COPD or asthma)
  2. serious mental illness (schizophrenia or bipolar disorder)
  3. anticipated to live in poverty and/or be homeless/underhoused

Exclusion Criteria:

* patients unable to provide informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Emotional Distress on the PROMIS-29 Profile c2.1 Scale | 3 months
  Measure of emotional distress as measured by anxiety and depression systems

SECONDARY OUTCOMES:
Social needs met | 3 months
  Number of social needs experienced by patients from a list (yes/no) at baseline and 3 month follow up
COVID related outcomes (patient-reported questionnaire built for this study) | 3 months
  Patient-reported COVID-related clinic or hospitalization visits and COVID vaccine status captured at baseline and 3 month follow up
Mortality related to COVID-19 and all cause mortality | 12 months
  Mortality (number of deaths) data obtained from administrative data source
Number of hospitalizations related to COVID-19 and all cause mortality | 12 months
  hospitalization (number of hospitalizations) data obtained from administrative data source

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No